CLINICAL TRIAL: NCT05600985
Title: Clinical Characteristics of Patients Developing Chronic Dry Eye After Refractive Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DED-RS
Record Dates: First submitted 2022-10-24; First posted 2022-11-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — basal tears
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DED after FS-LASIK: patients with dry eye disease (DED) after refractive surgery (RS）
  Interventions: Procedure: FS-LASIK
- DED without FS-LASIK: patients with dry eye who did not have refractive surgery
- normal control: subjects with no ocular symptoms and no previous ocular surgeries

INTERVENTIONS:
Procedure: FS-LASIK — Laser-assisted in situ keratomileusis, commonly referred to laser eye surgery or laser vision correction, is a type of refractive surgery for the correction of myopia, hypermetropia, and astigmatism.
  Other Names: Femtosecond laser-assisted in situ keratomileusis
  Groups: DED after FS-LASIK

SUMMARY:
In recent years, many scholars have studied the ocular surface damage of patients with dry eye disease（DED）after FS-LASIK, but there has been a lack of comprehensive observation and research on the relationship and difference between dry eye （DE）patients with and without LASIK. Therefore, the purpose of this study was to investigate the characteristics of ocular surface and cytokines after FS-LASIK, and further explain the pathogenesis of chronic dry eyes after FS-LASIK. In addition, we will also compare clinical characteristics and tear neuropeptide concentrations in patients with dry eye disease (DED) with and without chronic ocular pain following FS-LASIK, and to investigate correlations between ocular pain, clinical characteristics, and tear neuropeptide levels.

DETAILED DESCRIPTION:
A single visit cross-sectional study was performed. Approximately 40 chronic dry eye participants who had FS-LASIK more than 12month prior were recruited. Approximately 40 dry eye participants without refractive surgery history and 40 healthy participants without dry eye were also recruited as control groups. In addition, the patients with post-FS-LASIK DED were categorized into two groups based on the presence or absence of chronic ocular pain: (1) post-FS-LASIK DED patients with chronic ocular pain and (2) post-FS-LASIK DED patients without chronic ocular pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18years to 40 years
2. Male or female
3. DED patients based on Chinese Dry Eye Diagnosis Standard (2020) with or without FS-LASIK
4. Provision of written informed consent.

Exclusion Criteria:

1. active ocular infection, ocular inflammation, active ocular allergy, severe blepharitis or obvious inflammation of the eyelid margin, which in the judgment of the investigator may interfere with the interpretation of the study results.
2. Pregnant and lactating women, or those planning a pregnancy over the course of the study
3. Uncontrolled systemic disease
4. Suffer from diseases that may affect corneal nerves, such as keratoconus, trigeminal neuralgia, allergic conjunctivitis, etc.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients from Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-10-29 (Actual); Primary Completion 2023-09-18 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
ocular surface disease index (OSDI) | baseline
  OSDI is one of the most frequently used questionnaires for evaluation of dry eye
  . This includes 12 questions which measure the frequency of symptoms over the recent week, and the scores range from 0 to 100.
numerical rating scale (NRS) | baseline
  The NRS was used to evaluate ocular pain and consists of a numbered line from 0 to 10 scores that measures pain intensity: 0-1: no pain; 2-4: mild pain; 5-7: moderate pain; and 8-10: severe pain.
NPSI-Eye (range 0-100 score) | baseline
  Neuropathic Pain Symptom Inventory modified for the Eye (NPSI-Eye) (range 0-100 over a 24-hour recall period)
Tear break-up time (TBUT)(s) | baseline
  BUT is the time from normal blinking to the first appearance of a break in the tear film.
Corneal fluorescein staining (CFS) | baseline
  The degree of fluorescein staining of the cornea was evaluated using the National Eye Institute (NEI) scale of five corneal regions (central, superior, temporal, nasal, and inferior). The scores range from 0 to 15.

SECONDARY OUTCOMES:
the concentration of Interleukin-1β（IL-1β) (pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-1β levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-6 (IL-6) (pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-6 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-10 (IL-10) (pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-10 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-23 (IL-23) (pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-23 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-17A (IL-17A) (pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-17A levels will be quantified by Luminex immunoassay.
the concentration of tumor necrosis factor-α (TNF-α)(pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. TNF-α levels will be quantified by Luminex immunoassay.
the concentration of interferon-γ (IFN-γ)(pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IFN-γ levels will be quantified by Luminex immunoassay
the concentration of granulocyte-macrophage colony-stimulating factor (GM-CSF)(pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. GM-CSF levels will be quantified by Luminex immunoassay.
the concentration of substance P (SP)(pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. SP levels will be quantified by Luminex immunoassay.
the concentration of alpha-melanocyte-stimulating hormone (α-MSH) (pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. α-MSH levels will be quantified by Luminex immunoassay.
the concentration of β-endorphin (pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. β-endorphin levels will be quantified by Luminex immunoassay.
the concentration of neurotensin(pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. neurotensin levels will be quantified by Luminex immunoassay.
the concentration of oxytocin(pg/ml) | baseline
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. oxytocin levels will be quantified by Luminex immunoassay.
Schirmer Ⅰ test (SⅠt) (mm/5 minutes) | baseline
  The Schirmer I test is performed using sterile strips without anesthesia. The strips are placed in the lateral part of the inferior fornix of the eye for 5min and the extent of tear flow down was measured in millimeters.
tear meniscus height (TMH)(mm) | baseline
  The amounts of basal tears between the upper and lower eyelid margin.
Lissamine green staining | baseline
  To grade the temporal zone, the subject looks nasally; to grade the nasal zone the subject looks temporally. The upper and lower conjunctiva can also be graded.
meibomian gland dropout rate | baseline
  grade 0: no gland atrophy; grade 1: ≤1/3 gland atrophy; grade 2: 1/3 to 2/3 gland atrophy；grade 3: >2/3 gland atrophy.
corneal sensitivity (range, 60-0 mm) | baseline
  Corneal sensitivity will be measured in the right eye only using the Cochet-Bonnet aesthesiometer and the ascending method of limits to determine the threshold of stimulus detection.
sub-basal corneal nerve density (mm/mm2) | baseline
  Sub-basal corneal nerve plexus image will be acquired using a laser scanning confocal microscope.
Hamilton anxiety scale | baseline
  to evaluate the psychological status of patients. A total score of less than 7 indicates normal.
Hamilton Depression scale | baseline
  to evaluate the psychological status of patients. A total score of less than 7 indicates normal.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, M.D., Principal Investigator — Peking University Third Hospital; Lu Zhao, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao L, Zhou Y, Duan H, Zhang Y, Ma B, Yang T, Chen J, Chen Y, Qi H. Analysis of Clinical Characteristics and Neuropeptides in Patients with Dry Eye with and without Chronic Ocular Pain after FS-LASIK. Ophthalmol Ther. 2024 Mar;13(3):711-723. doi: 10.1007/s40123-023-00861-3. Epub 2024 Jan 8. PMID 38190027